CLINICAL TRIAL: NCT03567083
Title: STRENGTHS: Fostering Responsive Mental Health Systems in the Syrian Refugee Crisis - The Turkey Site
Brief Title: Implementation of Problem Management Plus (PM+) in Adult Syrian Refugees in Turkey: Pilot
Acronym: STRENGTHS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Sehir University (Other)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10/2017No:1
Record Dates: First submitted 2018-06-08; First posted 2018-06-25 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Anxiety; Depression; Posttraumatic Stress Disorder
Keywords: Refugees; Mental Health Problems
MeSH Terms: conditions — Anxiety Disorders; Depression; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E-CAU with Problem Management Plus (PM+) (Experimental): 30 participants will be randomly assigned to E-CAU with PM+ group. The PM+ is developed by the World Health Organization (WHO) especially for the communities who are exposed to adversity. PM+ (Dawson et al., 2015) belongs to a set of programs which are low-intensity, shorter, less expensive and trans-diagnostic (i.e., not condition-specific, but targeted at a broader set of symptoms of common mental disorders) programs to reduce common mental health symptoms (including depression, anxiety and stress symptoms) and improve psychosocial functioning.
  Interventions: Behavioral: Problem Management Plus (PM+)
- Enhanced care as usual (E-CAU) only (No Intervention): 30 participants will be randomly assigned to E-CAU group. CAU ranges from the free health services government provides to Refugee and Asylum Seekers Assistance and Solidarity Association's (RASASA) mental health services which are provided by the Psychological Support Unit (MHPSS Support Unit) which includes counselling as well. The enhanced care arm (CAU, with the addition of a referral document), is to be used as a benchmark for measuring the effectiveness of STRENGTHS's intervention, which is Problem Management Plus (PM+).

INTERVENTIONS:
Behavioral: Problem Management Plus (PM+) — This intervention is based on the WHO treatment guidelines for conditions related to stress (WHO, 2013). It is a 5-session intervention that is delivered by trained non-specialized workers or lay people, and is available in individual and group delivery formats for both children and adults. PM+ includes evidence-based techniques such as; problem solving, stress management, behavioral activation, and accessing social support. It has proved to be effective by two randomized controlled trials (RCTs) in Kenya and Pakistan (Bryant, Dawson, Schafer, Sijbrandij, & van Ommeren, 2016; Rahman, Hamdani, Awan, Bryant, Dawson, Khan, Mukhtar-ul-Haq Azeemi, et al., 2016).
  Arms: E-CAU with Problem Management Plus (PM+)

SUMMARY:
To implement Problem Management Plus (PM+) in Syrian refugees with this pilot study in Turkey with the aim of informing the definitive RCT about drop-out rates and estimated effect sizes.

DETAILED DESCRIPTION:
The STRENGTHS (Syrian REfuGees MeNTal HealTH Care Systems) study is a 5-year study that started in January 2017 with funding from the European Commission Horizon 2020 scheme and Turkey is one of the sites that this study will be conducted. The main aim of STRENGTHS in Turkey is to evaluate the feasibility, acceptability, effectiveness and cost-effectiveness of the culturally adapted psychological intervention Problem Management Plus (PM+) intervention for adult Syrian refugees in Turkey.

The current trial registration is for the pilot trial to investigate the feasibility and acceptability (e.g., obtain estimates of drop-out rates), to inform a full-scale, definitive randomized controlled trial. Study participants (n=60) will consist of adult Syrian refugees (18 years and older) in Turkey with self-reported functional impairment (WHODAS 2.0 >16) and elevated psychological distress (K10 >15.9). Participants will be randomly allocated either to the treatment group who will receive five sessions of PM+ or to the enhanced care-as-usual (E-CAU) group. Participants in the comparison group will receive E-CAU only. The primary outcome will be the decrease in psychological distress from baseline to three-month post-intervention assessment, measured through the Hopkins Symptoms Checklist (HSCL-25).

ELIGIBILITY:
Inclusion Criteria:

* Adults of 18 years or above
* Syrian under temporary protection status
* Arabic-speaking
* Elevated levels of psychological distress (K10 >15.9) and reduced psychosocial functioning (WHODAS 2.0 >16)

Exclusion Criteria:

* Acute medical conditions
* Imminent suicide risk or expressed acute needs/protection risks (e.g., a young woman who expresses that she is at acute risk of being assaulted or killed)
* Severe mental disorder (psychotic disorders, substance-dependence)
* Severe cognitive impairment (e.g., severe intellectual disability or dementia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2018-06-23 (Actual); Primary Completion 2019-01-21 (Actual); Study Completion 2019-01-21 (Actual)

PRIMARY OUTCOMES:
Hopkins Symptom Checklist-25 (HSCL-25) | Change from baseline assessment, at 1 week post-intervention assessment (6 weeks after baseline), and change from post-assessment at 3 month post-intervention assessment (4-4.5 months after baseline)
  The aim is to measure the change in psychological distress. Sub-scales can be calculated for depression (13 items) and anxiety symptoms (10 items). There are two items related to somatic symptoms. The items are rated on a 1-4 point Likert scale, with a well-validated cut-off score of 1.75. The current study will primarily look at the total score in which the lower values represent a better outcome. Furthermore, aim is to examine changes in caseness in depression, a cut-off score for the depression sub-scale of 2.1 will be used.

SECONDARY OUTCOMES:
PTSD Checklist for DSM-5 (PCL-5) | Change from baseline assessment, at 1 week post-intervention assessment (6 weeks after baseline), and change from post intervention assessment at 3 month post-intervention assessment (4-4.5 months after baseline)
  The aim is to measure the change in PTSD symptoms. PCL-5 is a 20-item checklist corresponding with the 20 DSM-5 PTSD symptoms. Items are rated on a 0-4 scale and add up to a total severity score of 80, with higher scores indicating worse symptomatology. The current study will primarily look at the total score in which the lower values represent a better outcome.
Psychological Outcome Measures (PSYCHLOPS) | Change from baseline assessment, at 1 week post-intervention assessment (6 weeks after baseline), and change from post intervention assessment at 3 month post-intervention assessment (4-4.5 months after baseline)
  The aim is to assess the change in self-identified problems. PSYCHLOPS consists of four questions. It contains three domains: 2 questions on problems, 1 question on function, and 1 question on well-being. Participants are asked to give free text responses to the problem and function domains. Responses are scored on a 0-5 scale producing a maximum score of 20 (six points per domain). The current study will primarily look at the total score in which the lower values represent a better outcome.
Client Service Receipt Inventory (CSRI) | Change from baseline assessment, at 1 week post-intervention assessment (6 weeks after baseline), and change from post-assessment at 3 month post-intervention assessment (4-4.5 months after baseline)
  The aim is to measure the change in the cost of care. CSRI was developed for the collection of data on service utilization, and related characteristics of people with mental disorders, as the basis for calculating the costs of care for mental health cost-effectiveness research. The current study will look at the change in the cost of care.
Access to health care: own questionnaire | Change from baseline assessment, at 1 week post-intervention assessment (6 weeks after baseline), and change from the post-intervention assessment at 3 month post-intervention assessment (4-4.5 months after baseline)
  The aim is to assess the change in access to health care. The questionnaire will include 70 questions on perceived access to health care. 57 of those questions will be two-way closed ended questions (yes or no) with the addition of the items "don't know" and "refused to answer". 13 of these questions are asking the type of help received (counselling/psychotherapy, psychological support, and medicines) with the addition of the items "don't know" and "refused to answer". The current study will look at the change in the access to health care.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Ceren Acartürk, Principal Investigator — Istanbul Sehir University
Locations (1):
- Refugee and Asylum Seekers Assistance and Solidarity Association's (RASASA), Istanbul, Sultanbeyli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The STRENGTHS project is consisted of various partners from different sites (such as the Netherlands, Jordan, Germany etc.). It is planned that the individual sites will be sharing their data with the researchers who are from these project partners. In addition to this, the partners will use the same Study Protocol while adapting it to their site.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The STRENGTHS project is a five year project which started in 2017. The individual participant data will be available for the other partners during the project which is between 2017 and 2022.
Access Criteria: The criteria for access is to be a partner of the STRENGTHS project.

REFERENCES:
- [Background] Dawson KS, Bryant RA, Harper M, Kuowei Tay A, Rahman A, Schafer A, van Ommeren M. Problem Management Plus (PM+): a WHO transdiagnostic psychological intervention for common mental health problems. World Psychiatry. 2015 Oct;14(3):354-7. doi: 10.1002/wps.20255. No abstract available. PMID 26407793
- [Background] Dawson KS, Schafer A, Anjuri D, Ndogoni L, Musyoki C, Sijbrandij M, van Ommeren M, Bryant RA. Feasibility trial of a scalable psychological intervention for women affected by urban adversity and gender-based violence in Nairobi. BMC Psychiatry. 2016 Nov 18;16(1):410. doi: 10.1186/s12888-016-1117-x. PMID 27863515
- [Background] Rahman A, Hamdani SU, Awan NR, Bryant RA, Dawson KS, Khan MF, Azeemi MM, Akhtar P, Nazir H, Chiumento A, Sijbrandij M, Wang D, Farooq S, van Ommeren M. Effect of a Multicomponent Behavioral Intervention in Adults Impaired by Psychological Distress in a Conflict-Affected Area of Pakistan: A Randomized Clinical Trial. JAMA. 2016 Dec 27;316(24):2609-2617. doi: 10.1001/jama.2016.17165. PMID 27837602
- [Derived] Acarturk C, Uygun E, Ilkkursun Z, Yurtbakan T, Kurt G, Adam-Troian J, Senay I, Bryant R, Cuijpers P, Kiselev N, McDaid D, Morina N, Nisanci Z, Park AL, Sijbrandij M, Ventevogel P, Fuhr DC. Group problem management plus (PM+) to decrease psychological distress among Syrian refugees in Turkey: a pilot randomised controlled trial. BMC Psychiatry. 2022 Jan 4;22(1):8. doi: 10.1186/s12888-021-03645-w. PMID 34983461